CLINICAL TRIAL: NCT04534335
Title: The SSSH's: SNOO Smart Sleeper Use in Post-Operative Infants With Congenital Heart
Brief Title: SNOO Smart Sleeper for Infants With CHD
Acronym: SHHH's
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Lori Erickson, Director, Remote Health Solutions, PhD, Children's Mercy Hospital Kansas City
Other Study IDs: STUDY00001376
Record Dates: First submitted 2020-08-27; First posted 2020-09-01 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Congenital Heart Disease; Infant Development; Technology
Keywords: Congenital Heart disease; Infant Sleep
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: SNOO Smart Sleep from Happiest Baby, Inc — Data related to the use of the SNOO itself (collected electronically) such as the amount of movement provided by the SNOO, etc., will be examined with the hemodynamic data obtained during the use of the SNOO. Clinical care data as it relates to the child will also be evaluated as it pertains to the use of the SNOO (this information will focus on the amount and frequency of narcotics administered to the infant). feasibility of use is the device intervention.

SUMMARY:
Study Title The SSSH Study: SNOO Smart Sleeper Use in Post-Operative Infants with Congenital Heart Disease is a single site, cross-sectional, feasibility study of an infant smart sleeper. The Primary Objective is to evaluate the feasibility of collecting and integrating clinical data and SNOO data. The secondary Objective(s) is To assess the feasibility of conducting a future broader trial by evaluating the parents willingness to give parental permission for participation in the use of the SNOO. Research Intervention(s)/ Investigational Agent(s) SNOO Smart Sleeper from Happiest Baby, Inc.There are approximately 300 new infants per year who undergo cardiac surgery at Children's Mercy Kansas City (CMKC) who are 6 months of age and 11kg or less at the time of surgery Sample Size. A maximum of 15 patients will be enrolled for this feasibility study over the study Duration for Individual Participant Length of hospitalization on 4Sutherland, average length of stay for this patient population is 30 days.

DETAILED DESCRIPTION:
Infants with congenital heart disease (CHD) are a low frequency but high acuity and stress population in the pediatric hospital setting. There are approximately 300 patients admitted a year that require cardiac surgery and are under the age of 6 months at Children's Mercy. These patients may spend less time in the hospital, but the care they require is often complex resulting in potential hemodynamic changes and pain responses for the infants. Smart technologies are used in CHD populations like single ventricle interstage monitoring at home, CHAMP App, but there are opportunities for baby-parent-nurse in-hospital smart solutions such as the SNOO Smart Sleeper bassinet by Happiest Baby INC . The SNOO Smart Sleeper has been used in more than 20 other hospitals across the country, including The University of Kansas Health System, mainly for infants related to preterm or neonatal abstinence syndrome (NAS). The SNOO utilizes some of the components of the 5 S's (swaddling, side/stomach position, shushing, swinging, and sucking) to aid as physical interventions for infant pain. This has been shown to be effective for pain reduction and less crying time after painful procedures . The calming response for infants has been seen to improve with soothing of the infant through supine mechanical movement, swaddling, and sound . A prospective observational cohort of preterm (32-36 weeks GA) neonates found that intermittent hypoxia and bradycardia significantly declined after use of womb-like soothing sound. The auditory neural pathways have close anatomical connection to the autonomic nervous system and the potential for auditory to parasympathetic response and reduced cardiac and respiratory rates are intriguing for evaluation in the infant population after cardiac surgery. The SNOO has yet to be used in the post-operative pediatric CHD population in the inpatient setting. The success in other fragile infant populations lends to a possible new area for use in the high risk CHD population in the post-operative recovery phase related to pain and hemodynamic changes.

ELIGIBILITY:
Inclusion Criteria:

* infants who have recently undergone cardiac surgery or cardiac catheterization for a stent for pulmonary blood flow at Children's Mercy Kansas City
* less than or equal to 6 months of age and under 11kg .

Exclusion Criteria:

* Greater than 6 months of age or over 11kg

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Only the families of patients that have already undergone a procedure for congenital heart disease will be approached for participation in this study. All female and male infants will qualify.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2022-05-28 (Actual); Study Completion 2022-09-12 (Actual)

PRIMARY OUTCOMES:
Length of time of utilization of SNOO for each infant | 6 months
  Feasibility of new device for use in the pediatric cardiac surgery infant population

SECONDARY OUTCOMES:
Number of parents receptive to use of the SNOO | 6 months
  Total number of parents consenting for feasibility trial

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Lysaught, BSN, MBA, Principal Investigator — Children's Mercy
Locations (1):
- Children's Mercy Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harrington JW, Logan S, Harwell C, Gardner J, Swingle J, McGuire E, Santos R. Effective analgesia using physical interventions for infant immunizations. Pediatrics. 2012 May;129(5):815-22. doi: 10.1542/peds.2011-1607. Epub 2012 Apr 16. PMID 22508924
- [Background] Moller EL, de Vente W, Rodenburg R. Infant crying and the calming response: Parental versus mechanical soothing using swaddling, sound, and movement. PLoS One. 2019 Apr 24;14(4):e0214548. doi: 10.1371/journal.pone.0214548. eCollection 2019. PMID 31017930
- [Background] Parga JJ, Bhatt RR, Kesavan K, Sim MS, Karp HN, Harper RM, Zeltzer L. A prospective observational cohort study of exposure to womb-like sounds to stabilize breathing and cardiovascular patterns in preterm neonates. J Matern Fetal Neonatal Med. 2018 Sep;31(17):2245-2251. doi: 10.1080/14767058.2017.1339269. Epub 2017 Jun 22. PMID 28587528
- See also: Happiest Baby, Inc 2020 — http://www.happiestbaby.com